CLINICAL TRIAL: NCT00069524
Title: Antihyperlipidemic Effects of Oyster Mushrooms
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001782-01 (NIH)
Record Dates: First submitted 2003-09-29; First posted 2003-10-01 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections; Hyperlipidemia
Keywords: Highly active antiretroviral therapy (HAART); Ritonavir; Oyster mushrooms; Non-HDL cholesterol; Complementary Therapies; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — pleurotolysin B, oyster mushroom

INTERVENTIONS:
Drug: oyster mushroom

SUMMARY:
The primary goal of this study is to evaluate the short-term safety and potential efficacy of oyster mushrooms (Pleurotus ostreatus) for treatment of hyperlipidemia in HIV-infected patients who are taking Kaletra, a protease inhibitor (PI) that is commonly used in highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
This is a single-arm, open-label, 8-week "proof of concept" pilot study in 20 subjects to determine if there are detectable lipid-lowering effects of oyster mushrooms in patients with HIV and hyperlipidemia who are taking Kaletra (a ritonavir-containing HAART regimen). The study will also assess whether the concurrent administration of oyster mushrooms and such regimens is safe, and investigate the mechanism of action whereby oyster mushrooms may exert their antihyperlipidemic effect.

ELIGIBILITY:
Inclusion criteria:

* Documented HIV infection (positive ELISA and Western Blot or measurable plasma HIV RNA).
* Taking Kaletra (ritonavir/lopinavir), a ritonavir-containing antiretroviral therapy, for at least 12 weeks
* Elevated non-HDL cholesterol >= 160 mg/dl as defined by the National Cholesterol Education Program guidelines (within 30 days of enrollment)
* AST or ALT <2.5 times the upper limit of normal (ULN) within 30 days of study entry.

Exclusion criteria:

* Currently receiving antihyperlipidemic treatment (e.g., statins, fibrates, bile sequestrants, niacin)
* Pregnancy or breastfeeding
* Documented history of myopathy or myalgias on HMG-CoA reductase inhibitors
* Documented history of rhabdomyolysis
* Documented diagnosis of diabetes mellitus
* Any condition that, in the judgment of the investigator, precludes successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-06; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- General Clinical Research Center, San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Abrams DI, Couey P, Shade SB, Kelly ME, Kamanu-Elias N, Stamets P. Antihyperlipidemic effects of Pleurotus ostreatus (oyster mushrooms) in HIV-infected individuals taking antiretroviral therapy. BMC Complement Altern Med. 2011 Aug 10;11:60. doi: 10.1186/1472-6882-11-60. PMID 21831304